CLINICAL TRIAL: NCT04032977
Title: A Multicenter, Double-blind, Randomized, Controlled Study of the Safety and Effectiveness of PN40082 for Lip Augmentation
Brief Title: Safety and Effectiveness of PN40082 for Lip Augmentation
Status: Completed | Type: Interventional
Sponsor: Prollenium Medical Technologies Inc. (Industry)
Collaborators: Symbio, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO 2018-02
Record Dates: First submitted 2019-07-19; First posted 2019-07-25 (Actual); Results first posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-05

CONDITIONS: Lip Augmentation

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, controlled, multicenter clinical study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only the unblinded treating investigator and unblinded assistant will be unblinded to the treatment. The remainder of study/site personnel remain blinded.
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (2):
- PN40082 (Experimental): Test device: PN40082 (manufactured by Prollenium Medical Technologies) is a clear, colorless gel in 1.0 mL pre-filled syringes with 25 mg/mL of stabilized hyaluronic acid and lidocaine 0.3% w/w
  Interventions: Device: PN40082; Device: Restylane Silk
- Restylane Silk (Active Comparator): Restylane Silk (manufactured by Q-Med AB for Medicis - A Division of Valeant Pharmaceuticals Corporation North America, LLC ) is a clear, colorless gel in 1.0 mL pre-filled syringes formulated to a concentration of 20 mg/mL of stabilized hyaluronic acid and lidocaine 0.3% w/w.
  Interventions: Device: PN40082; Device: Restylane Silk

INTERVENTIONS:
Device: PN40082 — To provide a 1-point improvement in the lip fullness grading scale score of subjects with very thin or thin lips or subjects with Fitzpatrick IV, V or VI to improve the LFGS score by 1 for 1 or both lips
Device: Restylane Silk — To provide a 1-point improvement in the lip fullness grading scale score of subjects with very thin or thin lips or subjects with Fitzpatrick IV, V or VI to improve the LFGS score by 1 for 1 or both lips

SUMMARY:
To compare the safety and efficacy profile of PN40082 versus Restylane Silk Injectable Gel with 0.3% lidocaine (Restylane Silk) for lip augmentation in approximately 158 subjects.

DETAILED DESCRIPTION:
The objective of the study is to compare the safety and efficacy profile of PN40082 versus Restylane Silk Injectable Gel with 0.3% lidocaine (Restylane Silk) for lip augmentation. Approximately 158 subjects will be randomized at approximately 7 sites in this is a double-blind, randomized, controlled, multicenter clinical study of subjects seeking lip augmentation. Subjects meeting inclusion/exclusion criteria will be randomized 1:1 to treatment with either PN40082 or Restylane Silk. The Evaluating Investigator will be blinded to the treatment. Injections of the study device will be performed by an unblinded Treating Investigator.

At each visit, the blinded Evaluating Investigator evaluations and subject evaluations of the treated areas will be performed and recorded. Visits and telephone contacts will occur at:

Visit 1 / Week 0 (Day 1) - baseline and treatment

* Day 3 (±2 days) - Safety follow-up telephone call
* Day 14 (±2 days) - Safety follow-up telephone call Visit 2 / Day 28 (±2 days) / Month 1 - interim visit (touch-up if necessary)
* Day 33 (±2 days) - Safety follow-up telephone call (for subjects with touch-up treatment
* Day 44 (±2 days) - Safety follow-up telephone call (for subjects with touch-up treatment) Visit 3 / Day 56 (±4 days) / Month 2 - interim visit Visit 4 / Day 84 (±4 days) / Month 3 - interim visit
* Day 112 (±4 days) / Month 4 - Safety follow-up telephone call
* Day 140 (±4 days) / Month 5 - Safety follow-up telephone call Visit 5 / Day 168 (±7 days) / Month 6 - End of Study (EOS) Visit. All subjects will undergo the consent procedure for the open label retreatment protocol.

Evaluations include:

Lip Fullness Grading Scale (LFGS) (Overall lip fullness considering both lips together, fullness of the upper lip and fullness of the lower lip) Perioral lines at rest severity scale (POL) (Overall perioral lines at rest severity considering both lips together, perioral lines at rest severity of the upper lip and perioral lines at rest severity of the lower lip) Patient Global Aesthetic Improvement (pGAI) Investigator Global Aesthetic Improvement (iGAI) Safety will be assessed by monitoring adverse events (AEs) at all study visits

Other Safety Evaluations include:

Lip Function Lip Sensation

Other evaluations include:

Investigator Ease of Use Assessment Swelling Assessment Subject Satisfaction with Lips Assessment Subjects participation will be approximately 6 months and the study is estimated to last 20 months from first subject first visit to last subject last visit.

ELIGIBILITY:
Inclusion Criteria:

1. Men or non-pregnant or non-breastfeeding women over 21 years of age
2. If female and of childbearing potential, a negative urine pregnancy test at Baseline (Day 1) and the subject agrees to use adequate contraception during the study period
3. Has an overall score of very thin, or thin on the LFGS, as agreed upon by the Treating and Evaluating Investigators, and desires at least a 1-point improvement in overall LFGS score; OR Has a Fitzpatrick skin phototype IV, V or VI and has an LFGS score of thick or full, as agreed upon by the Treating and Evaluating Investigators, and desires treatment to the vermilion body of 1 or both lips
4. Willing to give written informed consent

Exclusion Criteria:

1. Women who are pregnant, lactating, or planning a pregnancy
2. History of allergy, anaphylaxis or hypersensitivity to injectable hyaluronic acid products, local anesthetics of the amide type such as lidocaine, or to latex, or is planning to undergo desensitization therapy during the study
3. Has lip tattoos, piercings, facial hair, or scars that would interfere with visualization of the lips and perioral area for the effectiveness assessments
4. Has abnormal lip function, with inability to effectively sip water through a straw
5. Has abnormal lip sensation, with inability to feel a 0.4G monofilament or a cotton wisp at any site on the lip
6. Has moderate or severe abnormal lip asymmetry
7. Has any mass formation on the lip
8. Has dentures or any device covering all or part of the upper palate, and/or severe malocclusion or dentofacial or maxillofacial deformities as judged by the Treating Investigator. Subjects planning to undergo extensive dental procedures such as dental implants, multiple tooth extractions, or oral surgery should not participate. Minor dental procedures such as teeth cleaning and repair of caries are not exclusionary
9. Has undergone facial plastic surgery or received permanent facial implants (e.g., polymethylmethacrylate, silicone, polytetrafluoroethylene, polyacrylamide, lifting threads) anywhere in the face or neck, or is planning to be implanted with any of these products during the study
10. Has undergone semi-permanent dermal filler treatment (e.g., calcium hydroxylapatite, poly-L-lactic acid) in the lower face (below the orbital rim) within 12 months before enrollment or is planning to undergo such treatment during the study
11. Has undergone facial tissue augmentation with fat injections, botulinum toxin injections in the lower face (below the orbital rim), mesotherapy, or cosmetic procedures in the face or neck (e.g., face-lift, laser, photo-modulation, intense pulsed light, radio frequency, dermabrasion, moderate or greater depth chemical peel, microneedling, or other ablative procedures) within 9 months before enrollment or is planning to undergo any of these procedures during the study
12. Has used ANY lip filling agents within 12 months of study enrollment (hyaluronic acid products, collagen-based products, etc.)
13. Has used any lip plumping products or devices within 10 days before enrollment or is planning to use such products during the study
14. Has begun using any over-the-counter (OTC) or prescription oral or topical anti wrinkle products for the lips or around the mouth within 90 days before enrollment or is planning to begin using such products during the study (Subjects who have been on a stable regimen of such products for at least 90 days are eligible for the study and must continue their regimen throughout the study.)
15. Is on an ongoing regimen of anticoagulation therapy (e.g., warfarin), thrombolytics, or inhibitors of platelet aggregation or nonsteroidal anti inflammatory drugs (NSAIDs, e.g., aspirin, ibuprofen) or other substances known to increase coagulation time (e.g., herbal supplements with garlic or gingko) within 10 days of undergoing study device injections. Subjects who will withhold such therapy for 10 days before AND after any injection session may participate
16. Has a history or presence of bleeding disorders
17. Has used systemic corticosteroids or immunosuppressive medications within 30 days prior to treatment
18. Is on a concurrent regimen of lidocaine or structurally related local anesthetics (e.g., bupivacaine)
19. Has an active inflammation (skin eruptions such as cysts, pimples, rashes, or hives), infection, cancerous or precancerous lesion, or unhealed wound on the face
20. Has a history of known susceptibility to keloid formation or hypertrophic scars
21. Has porphyria
22. Has active herpes labialis lesions at the time of injections. Subjects with a history of herpes labialis who have had four (4) or more outbreaks in the 12 months prior to enrollment are also excluded even in the absence of lesions at the baseline visit
23. Has impaired cardiac conduction, severely impaired hepatic function, or severe renal dysfunction that, in the opinion of the investigator, would place them at risk of associated complications from these illnesses during the course of the study
24. Has any uncontrolled disease, i.e., a condition that has not been appropriately diagnosed, evaluated, and received medically appropriate treatment or care
25. Has severe cardiovascular disease; examples include but are not limited to New York Heart Association heart failure classification III or IV, unstable angina, and internal pacemakers. Potential subjects with other significant cardiovascular diseases should be discussed with the Medical Monitor before enrolling-

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2019-05-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Tennessee Clinical Research Center, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PN40082 | Restylane Silk
Started | 80 | 78
Completed | 71 | 70
Not Completed | 9 | 8
Not completed — Withdrawal by Subject | 6 | 1
Not completed — Lost to Follow-up | 2 | 7
Not completed — Pregnancy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PN40082 | Restylane Silk | Total
Number analyzed (Participants) | 80 | 78 | 158
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (11.85) | 49.2 (11.85) | 47.4 (11.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 76 | 156
  Male | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 18 | 44
  Not Hispanic or Latino | 54 | 60 | 114
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 15 | 27
  White | 65 | 61 | 126
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Overall Lip Fullness Grading Scale
Description: The Lip Fullness Grading Scale is a 5 point photonumeric rating scale with 0 being very thin lips (worse outcome) up to 4 being full lips (better outcome)
Time Frame: Visit 1 baseline to Visit 3 Month 2, 56 days
Population: Per-Protocol population is all randomized subjects who met all inclusion/exclusion criteria; received study device, completed Visit 5 within the specified window; had LFGS score by the Blinded Evaluating Investigator at Visit 3/Month 2 within the specified visit window, and had no significant protocol violations that would affect the treatment evaluation.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PN40082 | Restylane Silk
Number analyzed (Participants) | 54 | 55
score on a scale | 1.52 (.885) | 1.53 (.790)

2. Secondary Outcome: Treatment Success Lip Fullness Grading Scale
Description: Percent of subjects with Lip Fullness treatment success (responder: overall LFGS based on the Blinded Evaluating Investigator Assessment) at Visit 3/Month 2 where responder is defined as a subject with at least a 1-grade increase from baseline on the LFGS post augmentation The lip fullness grading scale is a 5 point photonumeric rating scale with 0 being very thin lips (worse outcome) to 4 being full lips (better outcome)
Time Frame: Visit 1 baseline to Visit 3 Month 2, 56 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PN40082 | Restylane Silk
Number analyzed (Participants) | 54 | 55
Participants | 49 | 51

3. Secondary Outcome: Treatment Success Perioral Lines Severity Scale
Description: Percent of responders with Perioral Lines Treatment Success overall on the POL severity scale at Visit 4/Month 3 (defined as a subject demonstrating ≥ 1-point improvement, i.e., decrease in severity, from baseline. The Perioral Lines at rest severity scale is a 4 point rating scale with 0 = None, a mouth with no perioral lines (better outcome) to 3 = Severe, being a mouth with many deep lines or crevices (worse outcome)
Time Frame: Visit 1 baseline to Visit 4 Month 3, 84 days
Population: Per Protocol population is all randomized subjects who met all inclusion/exclusion criteria; received study device, completed Visit 5 within the specified window; had LFGS score by the Blinded Evaluating Investigator at Visit 3/Month 2 within the specified visit window, and had no significant protocol violations that would affect the treatment evaluation. Of the per protocol population the subjects who had perioral injection at Visit 1 or Visit 2 and had POL assessed at Visit 4/Month 3
Measure: Count of Participants; unit: Participants
Arm/Group | PN40082 | Restylane Silk
Number analyzed (Participants) | 21 | 21
Participants | 14 | 12

4. Secondary Outcome: Change From Baseline to Visit 4/Month 3 in Overall Lip Fullness Grading Scale
Description: The lip fullness grading scale is a 5 point photonumeric rating scale with 0 being very thin lips (worse outcome) to 4 being full lips (better outcome)
Time Frame: Visit 1 baseline to Visit 4 Month 3, 84 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PN40082 | Restylane Silk
Number analyzed (Participants) | 54 | 55
score on a scale | 1.37 (.917) | 1.42 (.712)

5. Secondary Outcome: Change From Baseline to Visit 5/Month 6 in Overall Lip Fullness Grading Scale
Description: as for outcome 4
Time Frame: Visit 1 baseline to Visit 5 Month 6, 168 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PN40082 | Restylane Silk
Number analyzed (Participants) | 54 | 55
score on a scale | 1.00 (.727) | .93 (.634)

ADVERSE EVENTS:
Time Frame: Each subject was monitored for the occurrence of AEs, including serious adverse events (SAEs), starting immediately after the subject has signed the informed consent form (ICF). Each subject was followed for safety monitoring until he/she was discharged from the study, up to 6 months. No Follow-up procedures related to pregnancy, AEs, or SAEs continued beyond the end of the study, 6 months.
Arm/Group | PN40082 | Restylane Silk
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/78
Serious Adverse Events (participants affected / at risk) | 2/80 | 1/78
Other Adverse Events (participants affected / at risk) | 75/80 | 75/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PN40082 (N=80) | Restylane Silk (N=78)
Detached Retina Right Eye (Eye disorders) | 1 (1) | 0 (0)
Right Invasive Mammary Carcinoma, Stage 2 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Facial Paralysis (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PN40082 (N=80) | Restylane Silk (N=78)
Injection Site Bruising (General disorders) | 57 (57) | 44 (44)
Injection Site Erythema (General disorders) | 8 (8) | 8 (8)
Injection Site Mass (General disorders) | 6 (6) | 9 (9)
Injection Site Movement Impairment (General disorders) | 3 (3) | 6 (6)
Injection Site Pain (General disorders) | 17 (17) | 24 (24)
Injection Site Pruritus (General disorders) | 4 (4) | 3 (3)
Injection Site Swelling (General disorders) | 70 (70) | 70 (70)
Facial Asymmetry (Musculoskeletal and connective tissue disorders) | 12 (12) | 8 (8)
Headache (Nervous system disorders) | 1 (1) | 8 (8)

LIMITATIONS AND CAVEATS:
Due to blinded randomization, no men were randomized into the PN40082 group. Pooled analysis was provided to the FDA from previous studies to demonstrate safety in men.

Not enough subjects were randomized that required treatment of their perioral lines to demonstrate statistically non-inferiority.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-10-02): https://cdn.clinicaltrials.gov/large-docs/77/NCT04032977/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-09): https://cdn.clinicaltrials.gov/large-docs/77/NCT04032977/SAP_001.pdf